CLINICAL TRIAL: NCT07178171
Title: A Prospective, Single-Center, Exploratory Study of QL1706 Combined With Short-Cycle Anthracyclines or Taxanes for the Treatment of Early-Stage Triple-Negative Breast Cancer
Brief Title: A Study of QL1706 Combined With Short-Cycle Anthracyclines or Taxanes for the Treatment of Early-Stage TNBC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-Breast01
Record Dates: First submitted 2025-09-08; First posted 2025-09-17 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: TNBC, Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — pirarubicin; 130-nm albumin-bound paclitaxel; Carboplatin; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QL1706 combined with nab-paclitaxel and carboplatin (Experimental): QL1706, nab-paclitaxel and carboplatin
  Interventions: Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4); Drug: Nab-paclitaxel; Drug: Carboplatin (AUC 5)
- QL1706 combined with pirarubicin and cyclophosphamide (Experimental): QL1706, pirarubicin and cyclophosphamide
  Interventions: Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4); Drug: Pirarubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4) — QL1706
Drug: Pirarubicin — pirarubicin
  Arms: QL1706 combined with pirarubicin and cyclophosphamide
Drug: Nab-paclitaxel — nab-paclitaxel
  Arms: QL1706 combined with nab-paclitaxel and carboplatin
Drug: Carboplatin (AUC 5) — carboplatin
  Arms: QL1706 combined with nab-paclitaxel and carboplatin
Drug: Cyclophosphamide — cyclophosphamide
  Arms: QL1706 combined with pirarubicin and cyclophosphamide

SUMMARY:
Triple-negative breast cancer (TNBC) accounts for about 20% of breast cancers, is poorly differentiated, progresses rapidly, and frequently recurs, making it the subtype with the worst prognosis. Owing to the absence of actionable receptors on tumor cells, chemotherapy has historically been the mainstay of TNBC treatment.

With advances in basic research, more immune checkpoint inhibitors (ICIs) targeting distinct pathways have entered clinical use. Avellutolimab (QL1706) combines two engineered monoclonal antibodies-anti-PD-1 and anti-CTLA-4-in a fixed ~2:1 ratio. By blocking PD-1, it inhibits immune escape; by blocking CTLA-4, it relieves immune suppression and activates antitumor immunity. Preclinical studies show QL1706 has stronger antitumor activity than either anti-PD-1 or anti-CTLA-4 alone. Clinically, QL1706 monotherapy demonstrated notable efficacy as second-line therapy for advanced cervical cancer, with a median PFS of 5.4 months and manageable safety (2% discontinuation due to adverse events). Based on these data, QL1706 was approved in September 2024 for patients with recurrent or metastatic cervical cancer progressing after prior platinum-based therapy.

In the TNBC immunotherapy era, the optimal chemotherapy backbone remains uncertain, raising two key questions. First, with the introduction of immunotherapy-especially dual ICI regimens-can chemotherapy be de-escalated, and which patients are suitable for such de-escalation? Second, should anthracyclines be retained within immunotherapy-based regimens? The single-arm cTRIO study (ASCO 2023) used six cycles of paclitaxel plus carboplatin plus anti-PD-1 and achieved a pCR rate of 56.5%, despite enrolling patients with more advanced disease and higher nodal positivity. In contrast, translational analyses from NeoTENNIS (2024) suggest anthracyclines may promote immune activation and enhance the effects of immunotherapy. Consequently, small-sample exploratory clinical studies are needed to assess the feasibility of anthracycline-sparing chemotherapy strategies in the TNBC immunotherapy era.

For these reasons, we propose an exploratory neoadjuvant study in patients with early-stage TNBC using four cycles of QL1706 combined with either a taxane or an anthracycline. The study plans to enroll 30 patients with early-stage TNBC. Eligible patients will be randomized using a random number table into two cohorts for exploration: Cohort 1) QL1706 combined with nab-paclitaxel and carboplatin; Cohort 2) QL1706 combined with pirarubicin and cyclophosphamide. If a pCR is achieved, no further chemotherapy will be administered. If a pCR is not achieved, patients will subsequently receive four additional cycles of QL1706 plus pirarubicin and cyclophosphamide and four additional cycles of QL1706 plus nab-paclitaxel and carboplatin, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 and ≤70 years with newly diagnosed invasive breast cancer.
2. Triple-negative breast cancer (TNBC) with clinical stage cT2-T4 and cN0-cN3.
3. Unilateral disease.
4. No prior chemotherapy or immunotherapy for invasive breast cancer.
5. ECOG performance status of 0-1.
6. Adequate renal, hepatic, cardiovascular, and bone marrow function.
7. The patient voluntarily participates and signs the informed consent form.
8. According to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, patients should have measurable tumor lesion.
9. Estimated life expectancy ≥6 months
10. Female subjects enrolled must be surgically sterilized, postmenopausal, or agree to use at least one medically acceptable method of contraception (e.g., intrauterine device [IUD], oral contraceptives, or condoms) during study treatment and for 6 months after the end of study treatment. The serum or urine pregnancy test within 7 days prior to enrollment must be negative, and the subject must not be breastfeeding.
11. Able to comply with study and follow-up procedures and willing to adhere to the visit schedule and the prohibitions and restrictions specified in the protocol.

Exclusion Criteria:

1. History of invasive malignant tumor within ≤5 years prior to signing the informed consent form, except for adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix.
2. History of autoimmune disease;
3. Active hepatitis B or C virus infection, except for hepatitis B virus carriers or patients stabilized after antiviral therapy, who may be enrolled if HBV DNA titer is ≤500 IU/mL or <2500 copies/mL. Active hepatitis C is defined as known HCV antibody positivity with a known HCV RNA quantitative result above the lower limit of detection of the assay.
4. Presence of any active infection requiring systemic therapy.
5. Currently using corticosteroids or immunosuppressive agents.
6. Prior treatment with immune checkpoint inhibitors.
7. Presence of psychiatric disorders or other conditions that may affect patient compliance.
8. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
9. Pregnant or breastfeeding female patients.
10. Known allergy to the investigational drugs used in this study or their components.
11. Any other condition that, in the opinion of the investigator, makes the patient unsuitable for participation in this clinical trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
PCR rate | From first dose to surgery, approximately 12-16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be available upon reasonable request after publication of the main results. Data will be shared with qualified researchers with a methodologically sound proposal, subject to approval by the study steering committee.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after main publication; available for at least 5 years thereafter.
Access Criteria: Researchers may request access through the corresponding author by submitting a proposal and a data use agreement.